CLINICAL TRIAL: NCT04096664
Title: Efficiency and Acceptability of SIMEOX® Used Autonomously at Home for Bronchial Clearance in Patients With Cystic Fibrosis: Prospective, Randomized Controlled Study
Brief Title: Home Airway Clearance in CF Patients
Acronym: HomeCareSIMEOX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Physio-Assist (Industry)
Collaborators: Icadom (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Home-Care SIMEOX®
Record Dates: First submitted 2019-07-17; First posted 2019-09-20 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Pulmonary Cystic Fibrosis
Keywords: bronchial clearance; cystic fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Intervention Model Description: Adaptive prospective, randomized, controlled, multicenter trial, with hierarchical sequential analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SIMEOX (Experimental): Use the device for 3 months in addition to usual care
  Interventions: Device: SIMEOX
- Control (No Intervention): Usual care

INTERVENTIONS:
Device: SIMEOX — Use without obligation, in autonomous and at home of the bronchial clearance device: SIMEOX
  Arms: SIMEOX

SUMMARY:
Regular bronchial clearance is essential in patients with cystic fibrosis for their bronchial health. SIMEOX® (Physio-Assist, Aix en Provence, France) is an innovative medical device for the drainage of the bronchial tree.

By changing the rheological properties of mucus, SIMEOX® helps to mobilize secretions and assists their transport to the upper airways. This technology is based on fundamental research on bronchial mucus rheology. At the present time, SIMEOX® device is mainly used over a short period at the time or after an exacerbation in healthcare structures (hospitals, physiotherapy practices, post-care, and rehabilitation units, etc…). The clinical effects observed in the short term encourages long-term autonomous use by the patients themselves.

The overall objective of this study is to evaluate the efficiency and acceptability of SIMEOX® used at home by the patient himself for bronchial clearance in patients with cystic fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with Cystic fibrosis
* Stabilization of the disease, defined by an at least 4 weeks period since the end of an exacerbation, stabilization will be let to investigator's judgment.
* Age >12
* Requiring at least 1 bronchial clearing session each week (regardless of the technique)
* Patient (or patient's legal representative if applicable), capable to read and understand the procedure, and capable to express consent for the study protocol.

Exclusion Criteria:

* Severe pneumothorax or hemoptysis (more than 30ml per 24 hours) within 6 weeks before the inclusion day.
* Patient placed on a transplant waiting list
* Any contraindication to an instrumental bronchial clearance technique
* Patients already own and use SIMEOX at home
* Unavailable patient or patient wishing to move to a different region within three months after inclusion.
* Patient currently participating or having participated to another interventional clinical research within a month prior inclusion date, that may impact the study, this impact is left to the investigator's judgment.
* Persons referred by the French Public Health Code to Articles L1121-5 to L1121-8 (includes all protected persons: pregnant women (confirmed by measurement of the serum human chorionic gonadotropin level for any woman wishing to enter the protocol and under childbearing age < 60), parturient woman, breastfeeding mother, everyone deprived of his liberty by judicial or administrative decision, everyone subject to a legal protection measure.
* Initiation of treatment with a CFTR modulator within the last 3 months

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Respiratory score of CFQ-R questionnaire | Change from baseline at 3 months
  Relative variation in respiratory score of the CFQ-R questionnaire (Cystic Fibrosis Questionnaire -revised version) in the SIMEOX® treated group versus control group. Score range from 0 to 100, with higher score indicating better health.
Variation of forced expiratory volume in 1 second (FEV1) | Change from baseline at 3 months
  Relative variation of the forced expiratory volume in 1 second (FEV1) in the SIMEOX® treated group versus control group

SECONDARY OUTCOMES:
Total score of CFQ-R questionnaire | Change from baseline at 3 months
  Relative variation in the total score of the CFQ-R questionnaire (Cystic Fibrosis Questionnaire -revised version) in the SIMEOX® treated group versus control group.Score range from 0 to 100, with higher score indicating better health.
Safety of use assessed by incidence of Treatment-Emergent Adverse Events | During 3 months of use
  Take note and count all Treatment-Emergent Adverse Events to assess the safe use of SIMEOX® device autonomously at home
Satisfaction assessed by "Treatment Satisfaction Questionnaire for Medication"(TSQM) questionnaire | After 3 months of use
  Total score into a value ranging from the worst satisfaction 0 to the best satisfaction 100 of the TSQM questionnaire in the SIMEOX® treated group to assess the satisfaction
Acceptability assessed by the number of uses of SIMEOX® device | During 3 months of use
  Count the self-declared number of uses of the device SIMEOX by the patient in the SIMEOX® treated group to assess the acceptability of the device.
Pulmonary forced vital capacity (FVC) | Change from baseline at 3 months
  Relative variation of forced vital capacity in liter in the SIMEOX® treated group versus control group.
FEV1/ FVC ratio | Change from baseline at 3 months
  Relative variation of FEV1/ FVC ratio in % in the SIMEOX® treated group versus control group.
Forced expiratory flow | Change from baseline at 3 months
  Relative variation of forced expiratory flow in liter per second in the SIMEOX® treated group versus control group
Static lung compliance in Liter | Change from baseline at 3 months
  Relative variation of Static lung compliance in liter in the SIMEOX® treated group versus control group
Static lung compliance in % of predicted value | Change from baseline at 3 months
  Relative variation of Static lung compliance in % of predicted value in the SIMEOX® treated group versus control group
Airway resistance | Change from baseline at 3 months
  Relative variation of Airway resistance in cmH2O per liter per second in the SIMEOX® treated group versus control group
Diffusion capacity for carbon monoxide | Change from baseline at 3 months
  Relative variation of Diffusion capacity for carbon monoxide in % in the SIMEOX® treated group versus control group
Quality of life assessed by EQ-5D 5L questionnaire : a standardized instrument for measuring generic health status | Change from baseline at 3 months
  Relative variation of the scores of EQ-5D (a standardized instrument for measuring generic health status) questionnaire in the SIMEOX® treated group versus control group to asess the generic quality of life.Each 5 descriptive items have a value ranging from 1(best) to 5 (worst) and the visual analogic scale item should be scored from 0 (worst health) to 100 (best health).
Physical activity assessed by step counts and moderate-to-vigorous physical activity | Change from baseline at 3 months
  Compare the effect of SIMEOX autonomous treatment at home versus usual care on step counts and moderate-to-vigorous physical activity measured by actigraph device
Sleep quality assessed by sleep efficiency and fragmentation | Change from baseline at 3 months
  Compare the effect of SIMEOX autonomous treatment at home versus usual care on sleep efficiency and fragmentation measured by actigraph device
Fatigue assessed by VAS (visual analogue scale) | During 3 months of use
  Compare the effect of SIMEOX autonomous treatment at home versus usual care on fatigue experienced after a drainage session assessed by the VAS score between 0 and 10
Dyspnea assessed by mMRC (Modified Medical Research Council) score | Change from baseline at 3 months
  Compare the effect of SIMEOX autonomous treatment at home versus usual care on mMRC (Modified Medical Research Council) score into a value ranging from the least severe dyspnea 0 to the most serious dyspnea 4
Exacerbation rate | After 3 months of use
  Compare the effect of SIMEOX autonomous treatment at home versus usual care on respiratory exacerbation rate
First exacerbation | During 3 months of use
  Compare the effect of SIMEOX autonomous treatment at home versus usual care on the time to onset of the first exacerbation.
Hospitalization rate | After 3 months of use
  Compare the effect of SIMEOX autonomous treatment at home versus usual care on hospitalization rate for respiratory exacerbation
Hospitalization duration | After 3 months of use
  Compare the effect of SIMEOX autonomous treatment at home versus usual care on hospitalization duration for respiratory exacerbation
Antibiotic therapy | After 3 months of use
  Compare the effect of SIMEOX autonomous treatment at home versus usual care on antibiotic therapy rate (intravenous or oral)
Adherence telemonitoring feasibility | After 3 months of use
  Adherence telemonitoring feasibility is assessed by comparing self-declared data (number of treatment session) and electronically transmitted data. Electronically transmitted data will be transmitted by the SIMEOX-ANDROID application to an electronic secured platform.
  In the SIMEOX® treated group only.
Acceptability of SIMEOX-ANDROID application assessed by self-questionnaire AES (acceptability E-SCALE) | After 3 months of use
  Total score into a value ranging from the worst acceptability 6 to the best acceptability 30 of the self-questionnaire AES (acceptability E-SCALE) in the SIMEOX® treated group to assess the SIMEOX-ANDROID application acceptability

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Hamidfar, MD, Principal Investigator — CHUGA
Locations (20):
- France (20):
  - CHU Amiens Picardie, Amiens
  - CHU Angers, Angers
  - CHI Créteil, Créteil
  - Grenoble University Hospital : pneumo-pediatric department, Grenoble
  - Grenoble University-Affiliated Hospital : Pneumology department, Grenoble
  - CHU Lyon HCL, Lyon
  - Marseille University Hospital - Pneumology department, Marseille
  - Montpellier Hospital Center, Montpellier
  - Nice University-Affiliated Hospital : Pneumology department, Nice
  - Nice University-Affiliated Hospital : Pneumo-pediatric department, Nice
  - Hôpital Armand-Trousseau, Paris
  - Hôpital Robert Debré, Paris
  - CHU Reims, Reims
  - Fondation Ildys, Roscoff
  - CHU Felix Guyon, Saint-Denis
  - CHU De la Réunion Site SUD - Pôle Femme-Mère-Enfant, Saint-Pierre
  - CHU De la Réunion Site SUD, Saint-Pierre
  - CHU Toulouse - Hôpital Larrey, Toulouse
  - CHU Toulouse pediatric, Toulouse
  - Groupement Hospitalier Brocéliande Atlantique, Vannes

IPD SHARING:
Plan to Share IPD: No